CLINICAL TRIAL: NCT05758831
Title: A Prospective Randomized Trial of Non-inferiority Comparing RItuximab Versus Ocrelizumab in Relapsing-remitting Multiple Sclerosis
Brief Title: RItuximab Versus Ocrelizumab in Relapsing-remitting Multiple Sclerosis.
Acronym: TRIO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 35RC20_9812_TRIO
Record Dates: First submitted 2023-02-17; First posted 2023-03-07 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis; Relapsing-remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; Relapsing-remitting
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Intervention Model Description: multicenter, prospective, comparative (non inferiority), randomized, double blinded phase III/IV study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomisation code transmitted to the pharmacy preparing the treatment. Blind labelling of treatments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ocrelizumab (Active Comparator): Day 0 (300mg), Day 15(300mg), and then 300 mg every 6 months (M6, M12, M18 and M24)
  Interventions: Drug: Perfusion of treatment Ocrelizumab
- Rituximab (Experimental): Day 0 (1000mg), Day 15 (1000 mg), and then 500 mg every 6 months (M6, M12, M18 and M24)
  Interventions: Drug: Perfusion of treatment Rituximab

INTERVENTIONS:
Drug: Perfusion of treatment Rituximab — Perfusion of treatment (Mabthera®, Truxima®, Rixathon®, Ruxience®)
  Arms: Rituximab
Drug: Perfusion of treatment Ocrelizumab — Perfusion of treatment (Ocrevus®)
  Arms: Ocrelizumab

SUMMARY:
The goal of this randomized clinical trial is to compare relapse remitting multiple sclerosis (RRMS) patients treated by ocrelizumab or by rituximab followed for 2 years. The main question it aims to answer is : • to demonstrate the non-inferiority of rituximab versus ocrelizumab in active relapsing MS patients on the % of patients without disease activity at 2 years.

During the 2 years, the study includes 6 follow-up visits and the completion of various health and quality of life questionnaires. The protocol visits follow the usual schedule of treatment infusions for the disease (at initiation of treatment, 15 days after, and then every 6 months).

Two comparison groups: Researchers will compare rituximab treated patients versus ocrelizumab treated patients to see the % of patients without disease activity at 2 years.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is an autoimmune inflammatory disease of the central nervous system (CNS). This disease is the leading cause of non-traumatic disability in young adults and France is characterized by a high prevalence (currently 1/1000 inhabitants) of MS.

Clinical trials with B cell depleting therapies have shown efficacy in relapsing-remitting MS (RRMS) and are increasingly perceived as an important addition to the existing panel of Disease-modifying treatments (DMTs). Rituximab, a mouse chimeric anti CD20, is approved for non-Hodgkin's lymphoma, chronic lymphocytic leukemia, certain forms of vasculitis and Rheumatoid Arthritis with first marketing approval in 1998. Rituximab has undergone clinical testing in RRMS in 2008 in a phase II placebo-controlled trial, demonstrating the clinico-radiological efficacy in 104 patients. Despite these promising results and the absence of adverse events, its clinical development was interrupted by the manufacturer (Roche). However, for several years, rituximab has been increasingly prescribed (off-label) in Europe and USA in patients refractory to first-line therapies, with a very good safety and efficacy. Thus, rituximab is prescribed for 40% of RRMS patients treated in Sweden. Roche has then developed a humanized anti-CD20 monoclonal antibody (Ocrelizumab). Two phase III clinical trials (OPERA I and II) have demonstrated its efficacy in active RRMS. Ocrelizumab has just been authorized in France in this indication: RRMS patients with active disease (clinical or radiological). So, it can be prescribed as a first line or second line therapy in active RRMS patients.

According to literature, there are no biological arguments to think that ocrelizumab could be more effective in active RRMS compared to rituximab. Moreover, regarding safety, rituximab has been used for other indications for almost two decades and no serious concern has arisen.

The high cost of this new antibody (x6 to 10) compared to rituximab) makes it wonder about its place inside the anti-CD20 therapeutic strategy compared to rituximab for treating relapsing MS patients.

Hypothesis: Researchers hypothesize that rituximab and ocrelizumab have the same efficacy in active RRMS patients. Indeed, if the non-inferiority of rituximab on the % of patients without disease activity is confirmed by the trial, the potential medico-economic benefit from a societal perspective will be a strong argument to ask for authorization of rituximab in active RRMS.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting a relapsing remitting MS according to Mac Donald 2017 criteria, with clinical or radiological criteria of activity (ie at least one relapse AND/OR one new T2 lesion in the last 12 months before inclusion);
* Age between 18 and 55 years
* EDSS ≤ 5
* Brain MRI within 6 months before inclusion
* For women of childbearing potential*: effective contraception (effective contraception include oral contraception, intrauterine devices and other forms of contraception with failure rate <1%, for the duration of the study and until 12 months after last dose administered) * A woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.

A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.

* Having signed an informed consent form
* Patients covered with social insurance

Non-Inclusion Criteria:

* Secondary or primary progressive MS;
* Previous treatment by mitoxantrone, cladribine, alemtuzumab and anti CD20 therapies in the last two years;
* Previous treatment by fingolimod or natalizumab in the last 4 weeks;
* Treatment with high dose corticosteroids during the 30 days preceding the inclusion;
* Occurrence of a relapse less than 30 days before inclusion;
* Pregnancy or breastfeeding;
* Other neurologic or systemic disease;
* Concomitant participation or Participation in another therapeutic trial in the last 6 months;
* Incapacity to understand or sign the consent form;
* Contraindication to MRI;
* Contraindication to anti-CD20 therapies:

  * Receipt of a live or live-attenuated vaccine within 6 weeks prior to randomization
  * Active malignancy.
  * Any ongoing infection
  * Severe heart failure (New York Heart Association Class IV) or severe uncontrolled cardiac disease
  * Positive test for HIV, hepatitis B or C, or tuberculosis
  * Severe immune deficiency:
* Lymphopenia grade 3 (0.2 to 0.5 × 10^9/L) or higher grades
* Neutropenia grade 3 (0.5 to 1.0 × 10^9/L) or higher grades

  * Known hypersensitivity or other known side effects for any of the study medications, including co-medications such as high glucocorticosteroids
  * AST or ALT >=3ULN
  * Platelet (thrombocyte) count < 100 x 10^9/L
* Adults legally protected (under judicial protection, guardianship, or supervision), persons deprived of their liberty.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 386 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the non-inferiority of rituximab versus ocrelizumab in active relapsing MS patients on the percentage of patients without disease activity at 2 years. | at 2 years
  Percentage of patients without disease activity at 2 years (Disease activity is defined as:
  * At least one relapse between baseline and M24
  * OR MRI activity defined as Gd enhancing lesions at M6 or as the appearance of at least one new T2 lesion between M6 and M24)

SECONDARY OUTCOMES:
To compare the two groups (ocrelizumab vs rituximab) for Clinical Criteria : o Annualized relapse rate | at 2 years
  Relapses: annualized relapse rate
To compare the two groups (ocrelizumab vs rituximab) for Clinical Criteria : o Time of onset of the first relapse | at 2 years
  mean time of onset of the first relapse
To compare the two groups (ocrelizumab vs rituximab) for Clinical Criteria : o Percentage of patients without relapse | at 2 years
  Percentage of patients without relapse
To compare the two groups (ocrelizumab vs rituximab) for Clinical Criteria : o Percentage of patients without disability progression | at 2 years
  Percentage of patients without disability progression (Expanded Disability Status Scale-EDSS) (Disability progression will be defined as an increase of 1.5 pt if baseline EDSS=0, 1pt EDSS (if baseline 1 ≤ EDSS<6), or an increase of 0.5pt if baseline EDSS is ≥ 6; confirmed at 6 months.) EDSS : Minimum Score 1, Maximum score 10, higher scores mean a worse outcome.
MRI parameters : gadolinium (Gd) enhancing lesions | at 6 month
  - Mean number of Gd enhancing lesions at M6
MRI parameters : gadolinium (Gd) enhancing lesions | at 6 month
  - Percentage of patients with at least one Gd enhancing lesion(s)
MRI parameters : Mean Number of new T2 lesions | From Month 6 to Month 24
  - Mean number of new brain T2 lesions
MRI parameters : Percentage of patients with one or more new T2 lesions | From Month 6 to Month 24
  - Percentage of patients with one or more new brain T2 lesions
Patients quality of life : EQ-5D-5L | From baseline (Day 0) to every six month of follow up until Month 24
  Change in the EQ-5D-5L score
  The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
Patients quality of life : MusiQOL (Multiple Sclerosis International Quality of Life questionnaire) | From baseline (Day 0) to Month 12
  Change in the MusiQOL score
  The MusiQoL is a specific questionnaire comprising 31 questions describing nine dimensions of quality of life (Appendix 1):
  activities of daily living (eight items); psychological well-being (four); relationships with friends (four); symptoms (three); relationships with family (three); relationships with the health care system (three); emotional and sexual life (two); coping (two); rejection (two).
  Each item is scored from 1 (never/not at all) to 5 (always/very much). Before calculating the score of the dimensions, the scores of negatively written items are reversed. The score of a dimension is obtained by averaging the scores of its constituent items. The dimension scores are then transformed linearly into scores ranging from 0 to 100 (100 being the maximum quality of life level). A global quality of life score is also available.
Patients quality of life : MusiQOL | From baseline (Day 0) to Month 24
  Change in the MusiQOL score
  The MusiQoL is a specific questionnaire comprising 31 questions describing nine dimensions of quality of life (Appendix 1):
  activities of daily living (eight items); psychological well-being (four); relationships with friends (four); symptoms (three); relationships with family (three); relationships with the health care system (three); emotional and sexual life (two); coping (two); rejection (two).
  Each item is scored from 1 (never/not at all) to 5 (always/very much). Before calculating the score of the dimensions, the scores of negatively written items are reversed. The score of a dimension is obtained by averaging the scores of its constituent items. The dimension scores are then transformed linearly into scores ranging from 0 to 100 (100 being the maximum quality of life level). A global quality of life score is also available.
Patients experience : Musicare | From baseline (Day 0) to Month 12
  Change in the Musicare score
  Musicare is a questionnaire to assess the experience of both patients and caregivers of quality of care in MS, in accordance with psychometric standards. It comprises 35 items encompassing 5 domains: Information about the disease (11), Information about the treatments/medical investigation (8), Relationships with health care teams (8) Health care access (5) Reception in care structures (3).
  Each item is scored from 1 (Strongly agree) to 5 (Don't know).
Patients experience : Musicare | From baseline (Day 0) to Month 24
  Change in the Musicare score
  Musicare is a questionnaire to assess the experience of both patients and caregivers of quality of care in MS, in accordance with psychometric standards. It comprises 35 items encompassing 5 domains: Information about the disease (11), Information about the treatments/medical investigation (8), Relationships with health care teams (8) Health care access (5) Reception in care structures (3).
  Each item is scored from 1 (Strongly agree) to 5 (Don't know).
Medico-economic impact: cost-utility ratio, QALY | At 2 years
  Incremental Cost-Effectiveness Ratio (ICER) defined as the cost for QALY gained in "ocrelizumab group" versus "rituximab group" at 24 months.
Safety: Number of each adverse event | At 2 years
  Number of each adverse event will be compared between the two groups
Safety: Number of each severe adverse events | At 2 years
  Number of each severe adverse events will be compared between the two groups

CONTACTS AND LOCATIONS:
Locations (23):
- France (23):
  - Hospices Civils de Lyon Hôpital Neurologique Pierre Wertheimer, Lyon, Bron
  - CHRU de Brest - Hôpital la Cavale Blanche, Brest
  - Centre Hospitalier Universitaire de Caen, Caen
  - Centre Hospitalier de Pontoise - GHT NOVO, Cergy-Pontoise
  - Hôpital Gabriel Montpieds, Clermont-Ferrand
  - Centre hospitalier de Gonnesse, Gonesse
  - Groupe Hospitalier de l'Institut Catholique de Lille, Lille
  - Centre Hospitalier Universitaire de Limoges, Limoges
  - AP-HM - Hôpital la Timone, Marseille
  - CHRU de Montpellier - Hôpital Gui de Chauliac, Montpellier
  - Centre Hospitalier Régional de Nancy, Nancy
  - CHU de Nantes -Hôpital Nord Laennec, Nantes
  - CHU de Nice - Hôpital Pasteur 2, Nice
  - CHU de Nîmes - Hôpital Caremeau, Nîmes
  - AP-HP Höpital la Pitié-Salpétrière, Paris
  - Groupe Hospitalier Universitaire Henri Mondor, Paris
  - Hôpital Saint-Germain, Poissy
  - Centre Hospitalier de Cornouaille, Quimper
  - Centre Hospitalier Universitaire de Rennes, Hôpital Pontchaillou, Rennes
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen
  - CHRU de Strasbourg - Hôpital Hautpierre, Strasbourg
  - Hôpital Foch, Suresnes
  - CHU de Toulouse - Bâtiment Pierre Paul Riquet, Toulouse